CLINICAL TRIAL: NCT02097368
Title: Prospective Evaluation of Bulbar Function in Neuromuscular Patients
Brief Title: Bulbar Function in Neuromuscular Patients
Acronym: ORDEG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A00601-44
Record Dates: First submitted 2013-12-20; First posted 2014-03-27 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Neuromuscular Diseases
Keywords: Tongue strength; neuromuscular; swallowing
MeSH Terms: conditions — Neuromuscular Diseases | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- neuromuscular patient: Patients affected by neuromuscular pathology will be explored by tongue strength measurement, respiratory function measurement, swallowing tests and Magnetic resonance imaging
  Interventions: Procedure: tongue strength measurement; Procedure: respiratory function measurement; Procedure: swallowing tests; Other: Magnetic resonance imaging

INTERVENTIONS:
Procedure: tongue strength measurement — tongue strength measurement
Procedure: respiratory function measurement — respiratory function measurement
Procedure: swallowing tests — swallowing tests
Other: Magnetic resonance imaging — Magnetic resonance imaging

SUMMARY:
The main objective is prospectively study the upper airways function in an adult population of neuromuscular patients. The main measurement will be the evolution of tongue strength recorded each year during annual clinical evaluation on a 5 years period.

DETAILED DESCRIPTION:
The main objective is to study the function of the superior airways (tongue and pharynx) in an non invasive way in neuromuscular patients followed in the home ventilation unit of the Raymond POINCARE hospital (myopathy, neuropathy, disease of the neuromuscular junction or anterior horn) or of Necker Hospital and to detect prematurely the bulbar dysfunction.

The secondary objectives of this prospective monocentric observational physiopathological study are:

1. to study the correlation between the possible swallowing dysfunction and the anomalies of the respiratory parameters
2. to establish correlations between infraclinical or clinical and presence of morphological tongue anomalies detected by magnetic resonance imaging like in acid maltase deficiency.

The maximal tongue strength protrusion will be measured according to a method already used in the laboratory to explore sleep apnea syndromes.

Swallowing will be estimated by a non invasive method already used to highlight swallowing disorders in neurological and muscular pathologies This method will be associated with a method of recording of thoracic and abdominal movements.

Data wil be compared to a control database obtained for a previous study

ELIGIBILITY:
Inclusion Criteria:

* neuromuscular disorder
* age greater than or equal to 6
* Hospitalization in Home Ventilation Unit - Written informed consent

Exclusion Criteria:

* patient's refusal to participate
* major swallowing disfunction
* Acute respiratory failure
* no affiliation to social security

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients affected by neuromuscular pathology
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change of tongue strength measurement | 5 years
  Measurement using mechanical force transducer

SECONDARY OUTCOMES:
swallowing tests | 5 years
  Non invasive measurement of swallowing function using surface electromyography, accelerometry and inductance plethysmography
Respiratory parameters | 5 years
  Vital capacity and respiratory muscle strength measurement using spirometry and manometry
Vital capacity | 5 years
  Spirometry
Respiratory muscle strength | 5 years
  manometry (maximal inspiratory pressure and expiratory pressure)

CONTACTS AND LOCATIONS:
Overall Officials: David Orlikowski, MD, PhD, Principal Investigator — Centre d'Investigation Clinique et Technologique 805; Helene Prigent, MD,PhD, Principal Investigator — Centre d'Investigation Clinique et Technologique 805; Frederic Lofaso, MD, PhD, Principal Investigator — Centre d'Investigation Clinique et Technologique 805
Locations (2):
- France (2):
  - Home Ventilation Unit, Raymond Poincare Hospital, Garches
  - Non invasive ventilation Unit - Necker Hospital, Paris